CLINICAL TRIAL: NCT07293312
Title: Optimizing the Use of Virtual Reality in Rehabilitation for Individuals With Persistent Rotator Cuff-related Shoulder Pain
Brief Title: Optimizing the Use of Virtual Reality in Rehabilitation for Individuals With Persistent Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Full professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-3292
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Related Shoulder Pain
Keywords: Musculoskeletal Disorders; Virtual reality; Education; Shoulder; chronic pain intervention
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Masking Description: Participants will be blinded to the specific VR interventions they will perform to prevent anticipation or adjustment of their movements based on the intervention. For instance, they will not know whether their movements will be amplified or diminished compared to real-life motion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality interventions (Experimental): All participants will complete a four-week intervention, performing one of the four types of virtual reality (VR) exercises per week, so that each participant experiences all four exercises:
  1. Unimanual distraction task with normal visual feedback
  2. Bimanual distraction task with normal visual feedback
  3. Unimanual reaching task with augmented visual feedback
  4. Unimanual reaching task with diminished visual feedback
  During each session, participants will reach 18 targets positioned at heights of 60°, 90°, and 120° across three planes of motion (flexion, scaption, and abduction). Target positions will be adjusted to accommodate each participant's arm length and size. To ensure participant comfort, the session will end if repetitions are not completed within 2 minutes. The order of interventions will be randomized for each participant.
  Interventions: Other: Virtual reality unimanual distraction task; Other: Virtual reality bimanual distraction task; Other: Virtual reality unimanual reaching tasks with augmented visual feedback; Other: Virtual reality unimanual reaching tasks with decreased visual feedback

INTERVENTIONS:
Other: Virtual reality unimanual distraction task — Unimanual tasks (performed with the affected limb) with unaltered visual feedback will involve distraction exercises in which participants move a tray toward targets while keeping a ball balanced on the tray. Three trials with varying levels of friction between the ball and tray will be presented to manipulate the task's difficulty.
Other: Virtual reality bimanual distraction task — Bimanual tasks with unaltered visual feedback (targets positioned based on the affected limb) will involve distraction exercises in which participants move a tray toward targets while keeping a ball balanced on the tray. Three trials with varying levels of friction between the ball and tray will be presented to adjust task difficulty.
Other: Virtual reality unimanual reaching tasks with augmented visual feedback — Three trials with varying levels of visual feedback alteration will be performed, corresponding to a 0%, 25%, or 50% amplification of movement in the virtual environment compared to the real world. While virtual targets will appear farther apart, the actual movement required to reach them will remain the same across all trials.
Other: Virtual reality unimanual reaching tasks with decreased visual feedback — Three trials with varying levels of visual feedback alteration will be performed, corresponding to a 0%, 17%, or 33% reduction in movement in the virtual environment compared to the real world. Although the virtual targets will appear closer together, the actual movement required to reach them will remain the same across all trials.

SUMMARY:
The primary objective of this clinical trial is to investigate the effect of a block of four specific virtual reality (VR) exercises on upper limb function, pain, kinesiophobia, and pain catastrophizing in individuals with rotator cuff-related shoulder pain (RCRSP). The secondary objective is to examine participants' tolerability of different VR interventions.

Study Procedures:

Participants will:

* Attend a face-to-face assessment to confirm eligibility and receive a standardized pain neurophysiology education session (week 0).
* Visit the clinic once weekly for four weeks to undergo the VR interventions and review pain education concepts (Weeks 5 to 8).
* Complete online questionnaires evaluating upper limb function, kinesiophobia, pain, sense of presence, and cybersickness.

Interventions

Four VR interventions will be tested:

* Unimanual distraction task with normal visual feedback
* Bimanual distraction task with normal visual feedback
* Unimanual reaching task with augmented visual feedback
* Unimanual reaching task with diminished visual feedback

Findings will guide clinicians in selecting the most effective VR interventions for shoulder impairment and assess the feasibility of implementing VR in a private physiotherapy clinic for individuals with RCRSP.

DETAILED DESCRIPTION:
The use of virtual reality (VR) in rehabilitation has been shown to have positive effects on function and could enhance current rehabilitation interventions. However, the type of exercise to be performed, the specific added value of VR and the tolerance of the interventions performed remain poorly documented, which limits its clinical use. The primary objective of this project is to study the impact on function, pain, kinesiophobia and pain catastrophizing of a block of four specific VR exercises in individuals with chronic rotator cuff-related pain (RCRSP). The secondary objective is to examine participants' tolerance for different VR interventions.

Thirty adults with RCRSP will be recruited to participate in the study. Each participant will complete three assessment sessions: initial, pre-intervention, and post-intervention. The initial assessment will be conducted in person four weeks prior to the intervention to verify eligibility and provide standardized education on the neurophysiology of pain. This educational session aims to ensure a common level of understanding, improve adherence to the VR sessions, and facilitate the transfer of VR movements to daily activities.

The effect of the education will be assessed during the pre-intervention evaluation (week 4), conducted within seven days before the first VR session. The post-intervention evaluation (week 8), conducted within seven days following the 4-week intervention, will be used to address the study's primary objective. All questionnaires administered during the assessments and interventions will be completed online via REDCap.

The intervention will consist of four VR rehabilitation sessions, each involving a distinct type of task: 1)Unimanual distraction task with normal visual feedback; 2) Bimanual distraction task with normal visual feedback; 3) Unimanual reaching task with augmented visual feedback; and, 4) Unimanual reaching task with diminished visual feedback.

Outcome measures will include upper limb function, kinesiophobia, pain, participant satisfaction, sense of presence, and cybersickness.

To address the primary objective, repeated-measures ANOVAs will be conducted to compare outcomes across the three assessment time points (initial, pre-intervention [week 4], and post-intervention [week 8]). To address the secondary objective, repeated-measures ANOVAs will also be used to compare the effects of the different intervention types (unimanual vs. bimanual; augmented vs. diminished visual feedback).

This project will have an impact on both upper limb rehabilitation and the use of emerging VR technology in clinical settings. The project will provide a better understanding of the impact of VR intervention on symptoms, which is an important prerequisite for using VR in this population. It will also explore the type of intervention to be recommended in VR in complement to pain education.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff-related shoulder pain (screen by phone and then confirmed by the physiotherapist at the initial evaluation: pain over the deltoid and/or upper arm region, pain associated with arm movement [painful arc of movement], and familiar pain reproduced with loading or resisted testing during external rotation of the arm) for at least 6 months
* Minimum score of 15/100 on the shortened version of the Disabilities of the Arm, Shoulder, and Hand (1.5 times the minimally clinically important difference)

Exclusion Criteria:

* Unavailable for the 4 weeks intervention
* Cannot understand or read French
* Have a diagnosis of rheumatoid, inflammatory or neurodegenerative diseases
* Have received a corticosteroid injection or any other type of injection (e.g., platelet-rich plasma, prolotherapy, hyaluronic acid) in the past three months for their current condition
* Have bilateral shoulder pain
* Have pain in another upper limb joint
* Have signs of upper (e.g., bilateral paresthesia, hyperreflexia, or spasticity) or lower (e.g., decreased sensation or strength in dermatomes and myotomes, hypotonia, or hyporeflexia) motor neuron lesions
* History of shoulder surgery, dislocation, or fracture
* Presence of severe osteoarthritis, symptomatic acromioclavicular joint pathology, or adhesive capsulitis (defined as restriction of passive glenohumeral movement of at least 30% for two or more directions)
* Full thickness rotator cuff tear, identified by imaging or clinical tests (lag signs and gross weakness)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms and functional limitations specific to the upper limbs | post-intervention (week 8)
  The QuickDASH is an 11-item questionnaire, validated in individuals with rotator cuff-related shoulder pain, addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs. Higher scores indicate greater pain and functional limitations.

SECONDARY OUTCOMES:
Symptoms and functional limitations specific to the upper limbs | baseline
  The QuickDASH is an 11-item questionnaire, validated in individuals with rotator cuff-related shoulder pain, addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs. Higher scores indicate greater pain and functional limitations.
Symptoms and functional limitations specific to the upper limbs | pre-intervention (week 4)
  The QuickDASH is an 11-item questionnaire, validated in individuals with rotator cuff-related shoulder pain, addressing the level of difficulty in performing daily activities and the severity of the symptoms of the upper limbs. Higher scores indicate greater pain and functional limitations.
Functional limitations | baseline
  Functional limitations related to pain will be evaluated using the Pain Interference subscale of the Brief Pain Inventory (BPI). The Pain Interference subscale (7 items) measures the level of interference with function caused by pain on a scale from 0 to 10.
Functional limitations | pre-intervention (week 4)
  Functional limitations related to pain will be evaluated using the Pain Interference subscale of the Brief Pain Inventory (BPI). The Pain Interference subscale (7 items) measures the level of interference with function caused by pain on a scale from 0 to 10.
Functional limitations | post-intervention (week 8)
  Functional limitations related to pain will be evaluated using the Pain Interference subscale of the Brief Pain Inventory (BPI). The Pain Interference subscale (7 items) measures the level of interference with function caused by pain on a scale from 0 to 10.
Pain Severity | baseline
  Pain severity will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity from 0 to 10.
Pain Severity | pre-intervention (week 4)
  Pain severity will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity from 0 to 10.
Pain Severity | post-intervention (week 8)
  Pain severity will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity from 0 to 10.
Pain-related fear | baseline
  The Tampa Scale for Kinesiophobia will be used to evaluate pain-related fear. This scale is a 11-item scale designed to assess beliefs and behaviours associated with pain. Higher scores indicate a higher level of kinesiophobia.
Pain-related fear | pre-intervention (week 4)
  The Tampa Scale for Kinesiophobia will be used to evaluate pain-related fear. This scale is a 11-item scale designed to assess beliefs and behaviours associated with pain. Higher scores indicate a higher level of kinesiophobia.
Pain-related fear | post-intervention (week 8)
  The Tampa Scale for Kinesiophobia will be used to evaluate pain-related fear. This scale is a 11-item scale designed to assess beliefs and behaviours associated with pain. Higher scores indicate a higher level of kinesiophobia.
Pain catastrophizing | baseline
  The Pain Catastrophizing Scale will be used to evaluate pain catastrophizing. This scale is a 13-item scale designed to identify catastrophic thoughts about pain. Higher scores indicate a higher level of pain catastrophizing.
Pain catastrophizing | pre-intervention (week 4)
  The Pain Catastrophizing Scale will be used to evaluate pain catastrophizing. This scale is a 13-item scale designed to identify catastrophic thoughts about pain. Higher scores indicate a higher level of pain catastrophizing.
Pain catastrophizing | post-intervention (week 8)
  The Pain Catastrophizing Scale will be used to evaluate pain catastrophizing. This scale is a 13-item scale designed to identify catastrophic thoughts about pain. Higher scores indicate a higher level of pain catastrophizing.
Participants' satisfaction with their condition | baseline
  The Patient Acceptable Symptom State (PASS) will be used to assess participants' satisfaction with their condition. It asks patients whether they are satisfied with their current state and to rate their satisfaction on a 0-10 numeric scale.
Participants' satisfaction with their condition | pre-intervention (week 4)
  The Patient Acceptable Symptom State (PASS) will be used to assess participants' satisfaction with their condition. It asks patients whether they are satisfied with their current state and to rate their satisfaction on a 0-10 numeric scale.
Participants' satisfaction with their condition | post-intervention (week 8)
  The Patient Acceptable Symptom State (PASS) will be used to assess participants' satisfaction with their condition. It asks patients whether they are satisfied with their current state and to rate their satisfaction on a 0-10 numeric scale.
Pain severity related to the intervention | Immediately before, after and two days after each intervention (weeks 5 to 8)
  Pain severity related to the intervention will be evaluated using the Pain Severity subscale of the Brief Pain Inventory. The Pain Severity subscale of the BPI includes four items that measure pain intensity from 0 to 10.
Cybersickness | Immediately after each intervention (weeks 5 to 8)
  Cybersickness will be assess with the Simulator Sickness Questionnaire. This questionnaire contain questions about the intensity of symptoms related to the virtual reality intervention received.
Sense of presence | Immediately after each intervention (weeks 5 to 8)
  The Presence Questionnaire will be used to assess the sense of presence. This questionnaire contains questions about different aspects of the sense of presence with regard to the experienced virtual environment and the task being completed.
Satisfaction with interventions received | post-intervention (week 8)
  Participants will rate their satisfaction with treatment received ("not satisfied'', "satisfied'', "very much satisfied''), with the duration of treatments ("too short'', "long enough'', "too long''), with the frequency of treatments and with the time spent with the health professional during treatments ("not enough'', "just right'', "too much'') using a 3-item Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Mercier, OT,PhD, Study Director — Centre for Interdisciplinary Research in Rehabilitation and Social Integration (Cirris); Jean-Sébastien Roy, PT, PhD, Study Director — Centre for Interdisciplinary Research in Rehabilitation and Social Integration (Cirris)
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We are awaiting confirmation from the ethics research committee regarding permission to share individual participant data with other researchers. Once confirmed, we will outline the plan.